CLINICAL TRIAL: NCT03504644
Title: A Phase IB/II Study of Venetoclax (ABT-199) in Combination With Liposomal Vincristine or Vincristine Sulfate in Patients With Relapsed or Refractory T-Cell or B-Cell Acute Lymphoblastic Leukemia
Brief Title: Venetoclax and Vincristine in Treating Patients With Relapsed or Refractory T-cell or B-cell Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA9152; NCI-2017-01158 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA9152 (Other: ECOG-ACRIN Cancer Research Group); EA9152 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Adult Lymphoblastic Lymphoma; Recurrent B Acute Lymphoblastic Leukemia; Recurrent B Lymphoblastic Lymphoma; Recurrent T Acute Lymphoblastic Leukemia; Recurrent T Lymphoblastic Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory B Lymphoblastic Lymphoma; Refractory T Acute Lymphoblastic Leukemia; Refractory T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Specimen Handling; Spinal Puncture; Magnetic Resonance Spectroscopy; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ib (venetoclax, vincristine liposomal) (Experimental): Patients receive venetoclax PO QD on days 1-42 of cycle 1 and days 43-70 of cycle 2. Patients also receive vincristine liposomal IV over 1 hour weekly for 4 weeks starting on day 15 of cycle 1. Patients who achieve at least a stable disease response may continue treating at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the trial. Patients may also undergo CT and/or PET scan as well as a lumbar puncture as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Procedure: Positron Emission Tomography; Drug: Venetoclax; Drug: Vincristine Liposomal
- Phase II (venetoclax, vincristine liposomal/sulfate) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle. Patients also receive vincristine liposomal IV over 1 hour weekly for 4 weeks on day 1 of each cycle or vincristine sulfate IV weekly on days 1, 8, 15, and 22 of cycle 1 and once every 4 weeks on day 1 of each subsequent cycle. Cycles repeat every 28 days. Patients who achieve at least a stable disease response may continue treating at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the trial. Patients may also undergo CT and/or PET scan as well as a lumbar puncture as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Procedure: Positron Emission Tomography; Drug: Venetoclax; Drug: Vincristine Liposomal; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine Liposomal — Given IV
  Other Names: Lipid-Encapsulated Vincristine; Liposomal Vincristine; Onco TCS; Vincacine; VincaXome; Vincristine Liposome; Vincristine, Liposomal
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Phase II (venetoclax, vincristine liposomal/sulfate)

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of venetoclax and how well it works when given together with vincristine in treating patients with T-cell or B-cell acute lymphoblastic leukemia that has come back (recurrent) or does not respond to treatment (refractory). Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Chemotherapy drugs, such as vincristine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax together with vincristine may work better in treating patients with acute lymphoblastic leukemia compared to vincristine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of venetoclax in combination with vincristine liposomal (liposomal vincristine)/vincristine sulfate in patients with relapsed or refractory T-cell and B-cell acute lymphoblastic leukemia (ALL). (Phase I) II. Safety assessment and toxicity characterization after treatment of venetoclax in combination with liposomal vincristine in patients with relapsed or refractory T-cell and B-cell ALL. (Phase I) III. To determine the preliminary efficacy of venetoclax in combination with liposomal vincristine/vincristine sulfate to induce complete remission (CR)+ incomplete complete remission (CRi) in patients with relapsed or refractory T-cell and B-cell ALL. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the progression free survival, overall survival and toxicity after the combination treatment in patients with relapsed or refractory T-cell and B-cell ALL. (Phase II) II. To determine the rate of minimal residual disease (MRD) negativity rate of the combination. (Phase II)

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. To determine if genetic signature as determined by next generation sequencing can predict response to combination. (Phase II) II. To determine if immunophenotype of ALL is associated with response to combination. (Phase II) III. To determine if the BH3 profile is associated with response to combination. (Phase II) IV. To determine if relative expression of BCL-2 measure by flow cytometry is associated with response to combination. (Phase II)

OUTLINE: This is a phase Ib, dose-escalation study of venetoclax followed by a phase II study.

PHASE Ib: Patients receive venetoclax orally (PO) once daily (QD) on days 1-42 of cycle 1 and days 43-70 of cycle 2. Patients also receive vincristine liposomal intravenously (IV) over 1 hour weekly for 4 weeks starting on day 15 of cycle 1. Patients who achieve at least a stable disease response may continue treating at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the trial. Patients may also undergo computed tomography (CT) and/or positron emission tomography (PET) scan as well as a lumbar puncture as clinically indicated.

PHASE II: Patients receive venetoclax PO QD on days 1-28 of each cycle. Patients also receive vincristine liposomal IV over 1 hour weekly for 4 weeks on day 1 of each cycle or vincristine sulfate IV weekly on days 1, 8, 15, and 22 of cycle 1 and once every 4 weeks on day 1 of each subsequent cycle. Cycles repeat every 28 days. Patients who achieve at least a stable disease response may continue treating at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the trial. Patients may also undergo CT and/or PET scan as well as a lumbar puncture as clinically indicated.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 0: Patient must be considered a potential candidate for the trial

  * NOTE: Enrollment to Step 0 may occur prior to or following completion of the assessments to verify patient eligibility for Step 1 registration; bone marrow and/or peripheral blood specimens collected during Step 0 or prior to treatment on Step 1 must be submitted for central review in order for the patient to be considered evaluable; results will not be reported to the site and will not impact patient participation in the trial
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients must have a diagnosis of:

  * Relapsed or refractory B-cell or T-cell ALL after multi-agent chemotherapy
  * Patients with < 5% blasts may enroll on trial in phase I portion provided that minimal residual disease (MRD) is present at > 10^-3 as tested on an assay with minimum sensitivity of 10^-4 OR
  * Relapsed lymphoblastic lymphoma
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C): Age >= 18 years
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Adequate liver function with aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than 3 x upper limit of normal and total bilirubin less than 2 mg/dL within 10 days prior to first dose of study agent
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Circulating white blood cell (WBC) count must not be above 25 x 10^9/L at the time of registration

  * Patients with WBC count above 25 x 10^9/L are eligible if they have started steroids or hydroxyurea per institutional guidelines
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Glomerular filtration rate (GFR) of at least 40 mL/min within 7 days prior to first dose of study agent
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: All patients of childbearing potential must have a blood test or urine study with a minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG) within 2 weeks prior to registration to rule out pregnancy

  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients must not expect to conceive or father children by using accepted and highly effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 30 days after the last dose of venetoclax

  * Should a patient or a partner of a patient become pregnant or suspect they are pregnant while participating in the study, the treating physician should be notified immediately
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: No evidence of prior solid malignancy except adequately treated non-melanoma skin cancer, in situ cervical carcinoma, or any surgically- or radiation-cured malignancy continuously disease free for >= 2 years so as not to interfere with interpretation of radiographic response
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients may be enrolled with a prior allogeneic hematopoietic stem cell transplant (HSCT) but the transplant date must be at least 90 days before date of registration to step 1; patient must be off immunosuppression and without active graft versus host disease (GVHD) prior to registration to step 1 if previous HSCT
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 0: Patient must be considered a potential candidate for the trial

  * NOTE: Enrollment to Step 0 may occur prior to or following completion of the assessments to verify patient eligibility for Step 1 registration
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Relapsed or refractory B-cell or T-cell ALL, including lymphoblastic lymphoma, after at least one line of chemotherapy
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Age >= 18 years
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: ECOG performance status 0-2
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Adequate liver function with AST/ALT less than 3 x upper limit of normal and total bilirubin less than 2 mg/dL within 10 days prior to first dose of study agent
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Circulating WBC count must not be above 25 x 10^9/L at the time of registration to step 1

  * Patients with WBC count above 25 x 10^9/L are eligible if they have started steroids or hydroxyurea per institutional guidelines
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: GFR of at least 40 mL/min within 7 days prior to first dose of study agent
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: All patients of childbearing potential must have a blood test or urine study with a minimum sensitivity 25 IU/L or equivalent units of HCG within 2 weeks prior to registration to rule out pregnancy.

  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not expect to conceive or father children by using accepted and highly effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 30 days after the last dose of venetoclax

  * Should a patient or partner of a patient become pregnant or suspect she is pregnant while participating in this study, the treating physician should be informed immediately
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients may be enrolled with a prior allogeneic hematopoietic stem cell transplant (HSCT) but the transplant date must be at least 90 days before date of enrollment; patient must be off immunosuppression and without active GVHD prior to enrollment if previous HSCT. Low-dose steroids (10mg or less) are allowed

Exclusion Criteria:

* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients of childbearing potential must not be pregnant or breast-feeding due to risk of fetal harm by the chemotherapeutic agents prescribed in this protocol
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients with isolated testicular or central nervous system (CNS) relapsed disease are not eligible
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients must not have Burkitt's lymphoma/leukemia based on the World Health Organization (WHO) criteria
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients must not have active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF) or the use of CNS-directed local treatment for active disease within the prior 28 days; prophylactic intrathecal chemotherapy is allowed; previously treated CNS disease with documented clearance of the CSF will be allowed
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients will not be enrolled if they received prior chemotherapy within 2 weeks before registration to step 1 with the following exceptions: to reduce the circulating lymphoblast count or palliation or for ALL maintenance (mercaptopurine, methotrexate, vincristine, thioguanine, and/or tyrosine kinase inhibitors)
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients cannot have poorly controlled chronic viral infections including hepatitis B, C, or human immunodeficiency virus (HIV); HIV positive patients are allowed on this study if they have a CD4 count >= 400, and are on a stable antiviral regimen
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients with New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia may not be enrolled
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients with serious medical or psychiatric illness that in the opinion of the primary investigator is likely to interfere with study participation may not be enrolled
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients must not be taking any other experimental medications within 21 days prior to registration. Clinical trial medications that are Food and Drug Administration (FDA) approved will be allowed within 14 days prior to registration
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients should not have received the following within 7 days prior to the first dose of study drug:

  * Strong and moderate CYP3A inhibitors;
  * Strong and moderate CYP3A inducers
* ELIGIBILITY CRITERIA - PHASE I (ARMS A, B, C) - STEP 1: Patients must not have grade 3 or higher peripheral neuropathy or history of grade 3 or higher peripheral neuropathy. Patients with familial demyelinating disease like Charcot-Marie-Tooth disease are also excluded
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients with prior venetoclax treatment for ALL will be excluded
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not be pregnant or breast-feeding due to risk of fetal harm by the chemotherapeutic agents prescribed in this protocol
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: No evidence of prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical or breast carcinoma, or chemotherapy-surgically- or radiation-cured malignancy continuously disease free for >= 2 years
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients with isolated testicular or CNS relapsed disease are not eligible
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not have Burkitt's lymphoma/leukemia based on the WHO criteria
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not have active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF) or the use of CNS-directed local treatment for active disease within the prior 28 days; prophylactic intrathecal chemotherapy is allowed; previously treated CNS disease with documented clearance of the CSF will be allowed and once cleared, prophylactic intrathecal chemotherapy can be continued
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patient will not be enrolled if they received prior chemotherapy within 2 weeks before enrollment with the following exceptions: to reduce the circulating lymphoblast count or palliation (i.e., steroids or hydroxyurea), for ALL maintenance (mercaptopurine, methotrexate, vincristine, thioguanine, and/or tyrosine kinase inhibitors)
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients cannot have poorly controlled chronic viral infections including hepatitis B, C, or HIV; HIV positive patients with undetectable viral load are allowed
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients with NYHA class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia may not be enrolled
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients with serious medical or psychiatric illness that in the opinion of the primary investigator is likely to interfere with study participation may not be enrolled
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not be participating in any other clinical trial or taking any other experimental medications within 21 days prior to registration
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not have received the following within 7 days prior to the first dose of study drug or while on study treatment:

  * Strong and moderate CYP3A inhibitors;
  * Strong and moderate CYP3A inducers
* ELIGIBILITY CRITERIA - PHASE II (ARM D) - STEP 1: Patients must not have grade 3 or higher peripheral neuropathy or history of grade 3 peripheral neuropathy; patients with familial demyelinating diseases like Charcot-Marie-Tooth disease also excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of venetoclax (Phase I) | Up to 70 days
  Will be determined by dose limiting toxicity. The phase I portion of this study will use a standard 3+3 design.
Incidence of toxicities (Phase I) | Up to 5 years
  Toxicities will be assessed and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Complete remission (CR) + complete remission incomplete (CRi) rate (Phase II) | Up to end of cycle 3 (1 cycle = 28 days)
  A 90% confidence interval will be computed.

SECONDARY OUTCOMES:
Progression free survival (PFS) (Phase II) | From study registration to documented disease progression or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, and the median PFS along with its corresponding 95% confidence interval will be reported.
Overall survival (OS) (Phase II) | From study registration to death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, and the median OS along with its corresponding 95% confidence interval will be reported.
Incidence of toxicities (Phase II) | Up to 5 years
  Toxicity incidences will be assessed and graded according to the CTCAE and will be tabulated by patient cohort.
Change in intracellular BCL-2 expression (Phase II) | Baseline up to 5 years
  Will be assessed by flow cytometry and dichotomized into two groups by the median (low versus [vs] high). Univariate Cox proportional hazards (PH) models will be used to evaluate the association of the BCL-2 expression at baseline and immunophenotype (B-cell and T-cell acute lymphoblastic leukemia) with OS and PFS, separately. Logistic regression models will be used to investigate the association of the BCL-2 expression at baseline and immunophenotype with response (CR/CRi/partial remission [PR] vs others by 70 days). Multivariable Cox PH modelling and logistic regression modelling will also be used to adjust for the effect of covariates that are possibly associated with these efficacy outcomes.
Minimal residual disease (MRD) negativity rate (Phase II) | Up to 5 years

OTHER OUTCOMES:
Immunophenotype of acute lymphoblastic leukemia (Phase II) | Up to 5 years
  Logistic regression models will be used to investigate the association of the BCL-2 expression at baseline and immunophenotype with response (CR/CRi/PR vs. others by 70 days). Multivariable Cox PH modelling and logistic regression modelling will also be used to adjust for the effect of covariates that are possibly associated with these efficacy outcomes.
Genetic signature (Phase II) | Up to 5 years
  Will be assessed by next generation sequencing.
BH3 profile (Phase II) | Up to 5 years
  Will determine if the BH3 profile is associated with response to combination.
Expression of BCL-2 (Phase II) | Up to 5 years
  Will determine if relative expression of BCL-2 measure by flow cytometry is associated with response to combination.

CONTACTS AND LOCATIONS:
Overall Officials: Neil D Palmisiano, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (170):
- United States (163):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Palmisiano ND, Lee JW, Claxton DF, Paietta EM, Alkhateeb H, Park J, Podoltsev NA, Atallah EL, Schaar DG, Dinner SN, Webster JA, Luger SM, Litzow MR. A phase 1 trial of venetoclax in combination with liposomal vincristine in patients with relapsed or refractory B-cell or T-cell acute lymphoblastic leukemia: Results from the ECOG-ACRIN EA9152 protocol. EJHaem. 2024 Aug 8;5(5):951-956. doi: 10.1002/jha2.991. eCollection 2024 Oct. PMID 39415930